CLINICAL TRIAL: NCT04111770
Title: OPtimizaTIon of Left MAin PCI With IntravascuLar Ultrasound. The OPTIMAL Randomized Controlled Trial
Brief Title: The OPTIMAL Randomized Controlled Trial
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Philips Healthcare (Industry); Boston Scientific Corporation (Industry); Cardialysis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-013
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Left Main Coronary Artery Stenosis
Keywords: IVUS; PCI; Left Main; QCA; Treatment Strategy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVUS guided PCI (Experimental): Pre-procedural IVUS will be used to determine lesion characteristics and post-procedural IVUS to confirm correct implantation of stent.
  Interventions: Device: IVUS guided Percutaneous Coronary Intervention
- Angiography-guided PCI (Active Comparator): Qualitative or quantitative angiography will be used to determine lesion characteristics
  Interventions: Device: Qualitative or quantitative angiography will guide percutaneous coronary intervention

INTERVENTIONS:
Device: IVUS guided Percutaneous Coronary Intervention — Pre-procedural IVUS will be used to determine lesion characteristics and post-procedural IVUS to confirm correct implantation of stent.
  Arms: IVUS guided PCI
Device: Qualitative or quantitative angiography will guide percutaneous coronary intervention — Qualitative or quantitative angiography will be used to determine lesion characteristics
  Arms: Angiography-guided PCI

SUMMARY:
The OPTIMAL study is a randomized, controlled, multicentre, international study. A total of 800 patients will be randomized in a 1:1 fashion to Intravascular Ultrasound (IVUS)-guided PCI versus qualitative angio(QCA)-guided Percutaneous Coronary Intervention (PCI). Patients will be consented prior to the PCI procedure and then followed up to 2 years after the index procedure for the last enrolled patient. Patients will be followed-up at 1 month (telephone contact), 12 months (outpatient clinic visit or telephone call) and yearly after (outpatient clinic visit or telephone call).

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age;
2. De novo lesion in an unprotected left main coronary artery (ULMCA; ostial, shaft or distal) OR ostial left anterior descending artery (LAD) or ostial circumflex (LCX), both compatible with one Medina class of LM disease; or ostial intermediate branch disease;
3. PCI is considered appropriate and feasible by the treating interventionalist;
4. Silent ischemia, stable angina, unstable angina, or non-ST segment elevation MI;
5. Able to understand and provide informed consent and comply with all study procedures, including follow-up for at least 2 years.

Note: A patient with a prior CABG with no patent bypass on the left main coronary artery (LMCA) can be included.

Exclusion Criteria:

1. Patient is a woman who is pregnant or nursing;
2. Female patient of childbearing potential, i.e. who are not surgically sterile or post-menopausal (defined as no menses for 2 years without an alternative cause);
3. IVUS is strictly required for pre-PCI lesion severity assessment
4. ST-elevation myocardial infarction, cardiogenic shock;
5. Previous history of CABG with patent graft to the LAD and/or patent graft to the LCX;
6. Prior PCI of the LM, ostial LAD or ostial LCX at any time prior to enrollment;
7. Prior PCI of any other (i.e. non-LM, non-ostial-LAD and non-ostial-LCX) coronary artery lesions within 30 days prior to enrollment;
8. Patients unable to tolerate, obtain or comply with dual antiplatelet therapy for at least 6 months in stable patients and 1 year in ACS patients;
9. Known contraindication or hypersensitivity to everolimus, platinum-chromium, or to anticoagulants.
10. Patients requiring additional surgery (cardiac or non-cardiac) within 3 months post-enrollment;
11. Non-cardiac co-morbidities with a life expectancy less than 2 years;
12. Currently participating in another trial that is not yet at its primary endpoint. The patient is not allowed to participate in another investigational device or drug study for at least 12 months after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Patient-oriented Composite Endpoint (POCE) | 2-5 years follow up
  Patient-oriented Composite Endpoint (PoCE): composite of all-cause death, any stroke, any myocardial infarction (MI)*, any clinically indicated revascularization at longest follow-up.

SECONDARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 2-5 years follow up
  Device-oriented Composite Endpoint (DoCE) defined as the composite of: Cardiovascular death, target vessel MI, clinically indicated repeat revascularization of the target lesion at longest follow-up
Vessel-oriented Composite Endpoint (VoCE) | 2-5 years follow up
  Vessel-oriented Composite Endpoint (VoCE) defined as the composite of: left main related cardiac death, target vessel MI, clinically indicated -repeat revascularization of the left main vessels at longest follow-up.
Patient-oriented Composite Endpoint (POCE) | 2 year follow up
  Patient-oriented Composite Endpoint (PoCE): composite of all-cause death, any stroke, any myocardial infarction (MI)*, any clinically indicated revascularization at 2 years follow-up.
All individual components of PoCE at all time points. | 2-5 years follow-up
  All individual components of PoCE at all time points.
All individual components of DoCE at all time points. | 2-5 years follow-up
  All individual components of DoCE at all time points.
Definite and probable stent thrombosis | 2-5 years follow-up
  Definite and probable stent thrombosis according to ARC definition
Hospitalization for heart failure | 2-5 years follow-up
  Investigator reported hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Banning, Prof, Principal Investigator — Oxford University Hospitals NHS Trust; Luca Testa, Dr., Principal Investigator — Policlinco San Donato
Locations (28):
- Italy (8):
  - ASST Papa Giovanni XXIII, Bergamo
  - A.O.U. di Ferrara, Ferrara
  - Interventistica Cardiologica Strutturale, Florence
  - ASST Niguarda, Milan
  - Policlinco San Donato, Milan
  - Sant'Ambrogio Clinical Institute, Milan
  - Policlinico Umberto I, Rome
  - AOUI Verona, Verona
- Spain (10):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital de Bellvitge, Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital de Cabueñes, Gijón
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universiatrio V. Arrixaca, Murcia
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Clinico Lozano Blesa, Zaragoza
- United Kingdom (10):
  - Royal Victoria Hospital, Belfast
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex Country Hospital, Brighton
  - Bristol Royal infirmary, Bristol
  - University Hospital of Wales, Cardiff
  - Golden Jubilee National Hospital, Clydebank
  - Leeds General Infirmary, Leeds
  - St Bartholomew's Hospital, London
  - The Freeman Hospital, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Maria GL, Testa L, de la Torre Hernandez JM, Terentes-Printzios D, Emfietzoglou M, Scarsini R, Bedogni F, Spitzer E, Banning A. A multi-center, international, randomized, 2-year, parallel-group study to assess the superiority of IVUS-guided PCI versus qualitative angio-guided PCI in unprotected left main coronary artery (ULMCA) disease: Study protocol for OPTIMAL trial. PLoS One. 2022 Jan 7;17(1):e0260770. doi: 10.1371/journal.pone.0260770. eCollection 2022. PMID 34995276
- See also: Rationale and Design of the OPTIMAL Trial — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0260770